CLINICAL TRIAL: NCT06352866
Title: Phase II Trial of Siltuximab for Cytokine Release Syndrome Prophylaxis Prior to Treatment With Teclistamab in Relapsed or Refractory Multiple Myeloma (RRMM)
Brief Title: Siltuximab for Cytokine Release Syndrome Prophylaxis Prior to tx w/ Teclistamab in RRMM
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: Jack Khouri, MD (Other)
Responsible Party: Sponsor-Investigator, Jack Khouri, MD, Principal Investigator, MD, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE3A23
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma; Cytokine Release Syndrome; Refractory Multiple Myeloma; Immune Effector Cell Associated Neurotoxicity Syndrome
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Cytokine Release Syndrome | interventions — siltuximab

STUDY DESIGN:
Intervention Model Description: This study is an open label single cohort feasibility and efficacy study of siltuximab prophylaxis prior to infusion of teclistamab for treatment of RRMM. There is no planned dose escalation and no separate cohorts.
  Participants will receive a single dose of prophylactic siltuximab, 11 mg/kg, 2 hours prior to the administration of the first dose of teclistamab on day 1. There is no planned dose escalation of siltuximab, and teclistamab dosing will be done following the standard planned ramp-up. Participants will be hospitalized for 9 days according to teclistamab package insert and Cleveland Clinic institutional practice. Participants will be followed for the incidence of CRS and ICANS for the first two 22-day cycles of treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Siltuximab (Experimental): Participants will receive a single dose of prophylactic siltuximab, 11 mg/kg, 2 hours prior to the administration of the first dose of teclistamab on day 1. There is no planned dose escalation of siltuximab, and teclistamab dosing will be done following the standard planned ramp-up mentioned below. Participants will be hospitalized for 9 days according to teclistamab package insert and Cleveland Clinic institutional practice. Participants will be followed for the incidence of CRS and ICANS for the first two 22-day cycles of treatment.
  Interventions: Drug: Siltuximab; Drug: Teclistamab(FDA-approved)

INTERVENTIONS:
Drug: Siltuximab — Siltuximab is an investigational (experimental) drug that works by binding directly to human interleukin-6 (IL-6). IL-6 is a cytokine; these are products that are secreted by certain cells of the immune system and effect other cells in participant's body. IL-6 regulates immune, inflammatory and metabolic processes. Siltuximab has already been tested and approved for use by the FDA in participants with a condition called multicentric Castleman's disease, which is a disorder of the lymphatic system
Drug: Teclistamab(FDA-approved) — Teclistamab is a FDA-approved drug for the treatment of advanced MM after 4 lines of therapy.

SUMMARY:
The purpose of this study is to examine the safety, efficacy and feasibility of the use of one standard dose of siltuximab prior to teclistamab infusion. Siltuximab is an investigational (experimental) drug that works by binding directly to human interleukin-6 (IL-6). IL-6 is a cytokine; these are products that are secreted by certain cells of the immune system and effect other cells in participant's body. IL-6 regulates immune, inflammatory and metabolic processes. Siltuximab has already been tested and approved for use by the FDA in participants with a condition called multicentric Castleman's disease, which is a lymphoproliferative disorder. This study is being conducted to investigate if administration of a single dose of siltuximab will reduce the rates of and severity of Cytokine Release Syndrome (CRS) and Immune effector Cell-Associated Neurotoxicity Syndrome (ICANS) in participants prior to teclistamab administration. CRS and ICANS are adverse effects commonly experienced by participants being treated with teclistamab that are related to inflammation in the body. Siltuximab is experimental because it is not approved by the Food and Drug Administration (FDA) for prophylactic use prior to administration of teclistamab infusion.

DETAILED DESCRIPTION:
Cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity (ICANS) are clinically relevant toxicities of bsAbs and other T cell redirecting therapies. The armamentarium of immunotherapeutic approaches is expected to grow at exponential rates in the upcoming years, with an expansion of the diseases treated with this modality.

While the risk of CRS and ICANS is limited with most bsAbs(bispecific antibodies), these side effects can prevent a more widespread adoption of these therapies and impede their use in participants for whom access to tertiary or quaternary medical centers is limited.

The development of strategies that prevent CRS and ICANS occurring after bispecific antibodies can increase the prescription of these effective immunotherapies, in particular for participants for whom access to care is limited.

Siltuximab is a chimeric murine antibody that binds directly to IL-6 and has been used effectively in the treatment of CRS, with guidelines recommending its use in CRS cases refractory to tocilizumab.

Study hypothesis is that, through direct binding of IL-6, siltuximab can overcome the risk of increased IL-6 - mediated ICANS by decreasing the available IL-6 for blood brain barrier passage and by facilitating clearance of IL-6 through IL-6 receptor-mediated mechanisms.

Based on this rationale, a phase II study investigating the use of siltuximab for CRS and ICANS prophylaxis prior to therapy with the BCMAxCD3 bispecific antibody teclistamab.

This study will examine the safety, efficacy and feasibility of the use of standard doses of siltuximab prior to teclistamab infusion and will determine the rates of all grades as well as grade 2 or higher CRS and ICANS in participants given prophylaxis prior to teclistamab, which has well defined rates of CRS and ICANS. This will allow for a preliminary assessment of the efficacy of siltuximab as preventive measure against CRS and ICANS.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years of age and older.
2. Relapsed or refractory measurable multiple myeloma following prior treatment with ≥4 lines of anti-myeloma therapy slated for teclistamab monotherapy
3. Adequate bone marrow function including:

   * Hemoglobin ≥ 8g/dL (unless ≥50% bone marrow involvement by MM),
   * Absolute neutrophil count >1000 / µL (unless bone marrow involvement by MM)
   * Platelet count ≥30,000 / µL (unless bone marrow involvement by MM)
4. ECOG performance status 0 - 2
5. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year during the treatment period and for 3 months after the last dose of siltuximab.

   A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (< 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).

   Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.

   The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
6. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:

   1. With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period. Men must refrain from donating sperm during this same period.
   2. With pregnant female partners, men must remain abstinent or use a condom during the treatment period.

The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

1. Waldenström's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), or AL amyloidosis.
2. Known to be seropositive for human immunodeficiency virus or acquired immune deficiency syndrome.
3. Hepatitis B infection as defined according to the American Society of Clinical Oncology guidelines. In the event the infection status is unclear, quantitative levels are necessary to determine the infection status (Attachment 10). Hepatitis C (anti-hepatitis C virus [HCV] antibody positive or HCV-RNA quantitation positive) or known to have a history of hepatitis C. If positive, further testing of quantitative levels to rule out positivity is required.
4. Active central nervous system or meningeal involvement by MM.
5. Active bacterial, viral, fungal, mycobacterial, parasitic or other infection requiring systemic therapy within 2 weeks prior to first dose of study drug.
6. Active malignancy except for any of the following:

   * Adequately treated cutaneous basal cell carcinoma, squamous cell carcinoma, or in situ cervical cancer
   * Adequately treated Stage I cancer from which the subject is currently in remission and has been in remission for 2 years
   * Low-risk prostate cancer with Gleason score <7, prostate-specific antigen <10 ng/mL, and a stage of cancer at most cT2a, cN0, and CM0
   * Any other cancer from which the subject has been disease-free for ≥2 years
7. Participants with uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, pulmonary abnormalities or psychiatric illness/social situations that would limit compliance with study requirements.
8. Pregnant or breastfeeding women are excluded from this study because siltuximab therapy may be associated with the potential for teratogenic or abortifacient effects. Women of childbearing potential must have a negative serum pregnancy test. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with siltuximab, breastfeeding should be discontinued during treatment and for 3 months after the last dose of siltuximab. These potential risks may also apply to other agents used in this study.
9. Participants with history of clinically relevant and active CNS pathology such as epilepsy, seizure disorders, paresis, aphasia, uncontrolled cerebrovascular disease, severe brain injuries, dementia and Parkinson's disease.
10. Participants with history of severe hypersensitivity reaction to siltuximab or any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in CRS Rate | First two 22-day cycles after treatment initiation or until death, whichever occurs first.
  ASTCT criteria will be used to report CRS

SECONDARY OUTCOMES:
Safety assessment of a single dose of siltuximab as CRS prophylaxis | From the start of the infusion of the first dose of siltuximab until 22 days.
  Adverse events graded according to NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Incidence of grade ≥ 2 cytokine release syndrome after siltuximab prophylaxis | First two 22-day cycles after treatment initiation or until death, whichever occurs first.
  Response to siltuximab prophylaxis will be measured by incidence of all grade CRS and grade ≥ 2 CRS. Grading will be done according to the ASTCT consensus criteria
Incidence of all grade ICANS after siltuximab prophylaxis | First two 22-day cycles after treatment initiation or until death, whichever occurs first.
  Grading will be done according to the ASTCT consensus criteria
Incidence of adverse events after siltuximab prophylaxis | First two 22-day cycles after treatment initiation or until death, whichever occurs first
  Adverse events will be graded according to NCI CTCAE Version 5.0
Overall response rate | 6 months after treatment initiation or until disease progression, whichever comes first.
  Survival rates will be calculated using Kaplan Meier method
Progression free survival | 6 months after treatment initiation or until disease progression, whichever comes first.
  Survival rates will be calculated using Kaplan Meier method
Overall survival | 6 months after treatment initiation or until disease progression, whichever comes first.
  Survival rates will be calculated using Kaplan Meier method
Hospitalization rates | First two 22-day cycles after treatment initiation or until death, whichever occurs first
  Percentage as measured by Karnofsky Performance Scale to monitor hospitalization rates from 0 to 100, where 0 being death and 100 being normal, no complaints, no evidence of disease

CONTACTS AND LOCATIONS:
Overall Officials: Jack Khouri, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Center, Case Comprehensive Cancer Center Cleveland, Ohio
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Case Comprehensive Cancer Center Cleveland, Ohio, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Publications are expected to result from this trial. Individual participant data will not be shared.